CLINICAL TRIAL: NCT00071162
Title: Fibromyalgia Family Study Registry
Brief Title: Genetics of Fibromyalgia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sudha Iyengar, PhD, Case Western Reserve University
Other Study IDs: NIAMS-100
Record Dates: First submitted 2003-10-14; First posted 2003-10-15 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2009-03

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome; Chronic Fatigue Syndrome; Depression
Keywords: Pain; Fatigue; Sleep; Depression; Irritable Bowel Syndrome; Chronic Fatigue Syndrome
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Fatigue Syndrome, Chronic; Depression; Pain; Fatigue

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA, whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The Fibromyalgia Family Study identifies and collects blood samples from families with two or more members affected with Fibromyalgia Syndrome (FMS). The primary goal of the study is to identify genes that predispose people to FMS and/or symptoms related to FMS; identifying these genes may lead to a better understanding of the disease and more effective treatments.

DETAILED DESCRIPTION:
FMS predominantly affects women and is characterized by chronic widespread musculoskeletal pain, fatigue, sleep disturbance, and multiple tender points on physical examination. The pathophysiological mechanisms underlying FMS are not clearly understood, but neuroendocrine factors seem to be of major importance. Studies of familial association suggest that genetic factors play a role in FMS. This study will establish patterns of genetic linkage in families with FMS.

Participating family members will undergo a brief physical exam (including tender point exam), donate a blood sample, and complete a detailed questionnaire that includes experience with pain, fatigue, depression, bowel symptoms, headache, anxiety, and physical limitations. Measurements of serum serotonin and related compounds will also be obtained. To detect genetic factors, a genome-wide linkage scan using 405 microsatellite markers will be performed.

ELIGIBILITY:
Inclusion Criteria

* Diagnosed with fibromyalgia according to the criteria of the American College of Rheumatology
* Have at least one living family member who has also been diagnosed with fibromyalgia
* No other major rheumatological disease

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population of this study is family based and aimed to recruit 160 multic-case FMS families. We plan to perform a genome scan and evaluate 200-300 linkage markers to FMS and FMS-related traits. Future plans include establishing a DNA and data repository for distribution for future studies.
Sampling Method: Probability Sample
Enrollment: 560 (Actual)
Dates: Start 1999-09

CONTACTS AND LOCATIONS:
Overall Officials: Sudha Iyengar, PhD, Study Chair — Case Western Reserve University
Locations (4):
- United States (4):
  - University of Illinois at Peoria, Peoria, Illinois
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - University of Texas Health Sciences Center, San Antonio, Texas

REFERENCES:
- [Background] Yunus MB, Khan MA, Rawlings KK, Green JR, Olson JM, Shah S. Genetic linkage analysis of multicase families with fibromyalgia syndrome. J Rheumatol. 1999 Feb;26(2):408-12. PMID 9972977